CLINICAL TRIAL: NCT04312490
Title: Presentation, Patterns of Myocardial Damage, and Clinical Course of Viral Myocarditis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: Science and Technology Development Fund (STDF) (Unknown)
Responsible Party: Principal Investigator, Ayman khairy Mohamed, assistant professor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 26393
Record Dates: First submitted 2020-03-11; First posted 2020-03-18 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Myocarditis Viral
Keywords: VIRAL MYOCARDITIS

STUDY DESIGN:
Intervention Model Description: Prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients (Experimental): all patients with myocarditis
  Interventions: Diagnostic Test: endomyocardial biopsy

INTERVENTIONS:
Diagnostic Test: endomyocardial biopsy — Endomyocardial biopsies will be stained with Masson's trichrome as well as Giemsa and examined by light microscopy. For immunohistology, tissue sections will be treated with an avidin-biotinimmunoperoxidase method (Vectastain-Elite ABC Kit, Vector, Burlingame, Calif), with application of the following monoclonal antibodies: CD3 (T cells; Novocastra Laboratories, Newcastle, UK), CD68 (macrophages, natural killer cells; DAKO, Hamburg, Germany), and HLA-DR-α (DAKO, Hamburg, Germany
  Other Names: Quantitative real-time PCR; Restriction fragment length polymorphism-PCR for B19V genotyping; Histological and Immunohistochemistry analysis

SUMMARY:
Viral myocarditis has been recognized as a cause of congestive heart failure, however diagnosis and treatment represents a challenging process. Recently, there is an increasing frequency of different cardiotropic viruses in the clinical setting of myocarditis. The introduction of the new molecular techniques in analysing the etiologic agent of acute myocarditis has enhanced significantly the knowledge on the molecular epidemiology of these viruses. The etiology of patients admitted to our university hospital remains unclear. It is therefore important to identify the aetiology associated with myocardial infections.

The purpose of the present study is to analyze the prevalence of a broad spectrum of cardiotropic viruses, including enteroviruses, adenoviruses and parvo B19 virus, in adults with suspected myocarditis with special reference to B19 virus due to its increasing prevalence nowadays.

The results of this study will provide a very important information for the prevalent infectious viral agents in our university hospital which will guide treatment protocol.

DETAILED DESCRIPTION:
Objectives

1. There are almost no data regarding the relative prevalence of viral pathogens associated with myocarditis and the demographic and clinical features related to these infections in Egypt. Therefore, our main interest is to determine the prevalence of the most common viruses in clinically relevant (i.e., hospitalization- requiring) patients with acute or chronic myocarditis, using highly sensitive molecular techniques as the diagnostic tool.
2. Our second aim is to determine the distribution of mono- and coinfections between these viral agents.
3. Finally, to correlate between the microbiological findings in this study and patient characteristics including age, sex, clinical features, regional distribution, and degree of urbanization (determined on the basis of the size of the city and the density of the population) of the patients.

ELIGIBILITY:
Inclusion Criteria:

* all patients with recent unexplained heart failure in last 3 months and diagnosed as myocarditis by cardiac magnetic resonance (CMR) after exclusion of ischemic (by coronary angio) or valvular (by detailed ECHO) causes.

Exclusion Criteria:

* ischemic cardiomyopathy.
* peripartum cardiomyopathy
* valvular etiology of heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
prevalence of the most common viruses | 12 months
  our main interest is to determine the prevalence of the most common viruses in clinically relevant (i.e., hospitalization- requiring) patients with acute or chronic myocarditis, using highly sensitive molecular techniques as the diagnostic tool.

SECONDARY OUTCOMES:
Determine the distribution of mono- and co-infections between these viral agents. | 12 months
  Using PCR techniques to detect if single infection or multiple viral infection per pateint

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hassan AKM, Fouad DA, Refaiy A. Demographic features and prevalence of myocarditis in patients undergoing transarterial endomyocardial biopsy for unexplained cardiomyopathy. Egypt Heart J. 2017 Mar;69(1):29-35. doi: 10.1016/j.ehj.2016.09.005. Epub 2016 Oct 10. PMID 29622952
- [Derived] Khidr SS, El-Mokhtar MA, Asaad SR, Hetta HF, Abdel-Rahim MH, Youssef AAA, Hassan AKM. Clinical course, viral etiology, and the diagnostic workup for patients with suspected myocarditis: a single-center prospective study. BMC Cardiovasc Disord. 2022 Sep 6;22(1):396. doi: 10.1186/s12872-022-02833-0. PMID 36068503